CLINICAL TRIAL: NCT03688633
Title: Pilot Study, Single-blind, Candesartan Versus Usual Care of Peripheral Neuropathy Development Induced by Vincristine (PNIV) in Patients Treated for Lymphoma B
Brief Title: Candesartan in Peripheral Neuropathy
Acronym: NEUPERSART
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Patient Recruitment Failure
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: I16016 /NEUPERSART; NCT03805867 (obsolete NCT alias)
Record Dates: First submitted 2018-09-08; First posted 2018-09-28 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-09

CONDITIONS: Peripheral Neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases | interventions — candesartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Candesartan (Experimental)
  Interventions: Drug: Candesartan
- Usual care (Active Comparator)
  Interventions: Other: Usual care

INTERVENTIONS:
Drug: Candesartan — Candesartan treatment with dose adjustments (8-16mg/day) during 6 months in accordance with adverse effects
  Arms: Candesartan
Other: Usual care — patients will be followed as usual
  Arms: Usual care

SUMMARY:
Background:

Chemotherapy induced peripheral neuropathy (CIPN) is often painful, and is caused by neurotoxic chemotherapy including vincristine. It is a cause of significant impairment in quality of life in patients surviving to a solid cancer or malignant lymphoma. The only recognized prevention is based on pre-existing neuropathy and early detection of neuropathic signs and symptoms in individuals subjected to neurotoxic chemotherapy, justifying sometimes a change in the therapeutic strategy when other molecules are available. It seems obvious that to identify early markers of CIPN and to develop preventive therapeutic strategies, are priorities for improving patients' quality of life and enable them to follow optimal treatment.

Purpose:

To describe in patients treated for non-Hodgkin's type B malignant lymphoma with multidrug therapy containing vincristine, the impact of candesartan on the occurrence of neuropathy measured by the variation of TNSc (Total Neuropathy Score clinical version, evaluating clinical signs of neuropathy)

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and over and to be treated with Vincristine for non-Hodgkin B lymphoma (first line treatment)
* All the patients have to be treated with the same chemotherapy protocol (CHOP with or without Rituximab) to avoid confounding factors
* Normal renal function as measured by CKD-EPI > 30 mmol / min / 1.73 m2
* Serum potassium < 5.5 mmol / l
* Systolic arterial pressure > 100 mm Hg (lying and standing position)
* affiliated with a social security
* For women of childbearing age: under "highly effective" contraception and negative pregnancy test at inclusion. Highly effective contraception:

  * Combined hormonal contraceptive (containing estrogen and progesterone) (oral, intravaginal, or transdermal) or only progesterone (oral, injectable or implantable),

Exclusion Criteria:

* Patients with pre-existing neuropathy, Chronic ethylism, HIV infection, etc.
* Patients under guardianship or unable for another reason to give informed consent.
* Intolerance to sartans
* Intolerance to excipients : galactose , lactose.
* Patients already treated with ACE inhibitors, ARBs or/and diuretics sparing

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-05-27 (Actual)

PRIMARY OUTCOMES:
TNSc score variation between V1 and V4 | Between the base time (V1) and the end of chemotherapy (15 week later).
  The primary endpoint in this clinical study is the V1 - V4 variation of the TNSc score TNSc is the Total Neuropathy Score Clinical version scale
  Validated 7-item TNSc quantifies subjective sensory and motor symptoms, vibration sensation, strength, and reflexes.Items are rated using a 0 to 4 scale and summed to obtain a total score ranging from 0 to 28. Higher scores reflect more severe neuropathy.
  The evaluation of the TNSc will be performed by a blinded evaluator of the randomization group

SECONDARY OUTCOMES:
TNSc score variation between V1 and V3 | Between the base time (V1) and V3 (9 week later)
  VariationVariation between V1 and V3 of the TNSc score. TNSc is the Total Neuropathy Score Clinical version scale
  Validated 7-item TNSc quantifies subjective sensory and motor symptoms, vibration sensation, strength, and reflexes.Items are rated using a 0 to 4 scale and summed to obtain a total score ranging from 0 to 28. Higher scores reflect more severe neuropathy.
  The evaluation of the TNSc will be performed by a blinded evaluator of the randomization group.
Variation of visual analog scale (VAS) | Between the base time (V1) and 9 week and 15 week later
  Variation oh the VAS score between V1 - V3 and between V1- V4 The visual analogue scale (VAS) is commonly used as the outcome measure to characterize the intensity of pain . It is presented as a 100-mm horizontal line on which the patient's pain intensity is represented by a point between the extremes of "no pain at all" and "worst pain imaginable."
  Higher scores reflect more severe pain.
Adverse effects | At baseline and each cycle up to 16 week
  any adverse/ side effect will be evaluated

OTHER OUTCOMES:
Lipid peroxidation | through study completion, an average of 2 years
  Theses markers of vincristine-induced axonal involvement Lipid peroxidation will be assessed by measurement of MDA malondialdehyde (TBARS) and 8-Isoprostane
Oxidative stres | through study completion, an average of 2 years
  Oxidative stress will be evaluated by measuring the activities of superoxide dismutase (SOD) and glutathione peroxidase (GHS-PX).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Limoges, Limoges, France

IPD SHARING:
Plan to Share IPD: No